CLINICAL TRIAL: NCT00295659
Title: What is the Optimal Method for Screening and Diagnosis of Gestational Diabetes? An RCT to Evaluate Incidence, Cost-Effectiveness and Clinical Outcomes Using Three Methods
Brief Title: An RCT to Evaluate Incidence, Cost and Clinical Outcomes Using 75 vs 100g. Screening Methods for Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: Canadian Diabetes Association (Other)
Other Study IDs: CDA 200665
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2005-09

CONDITIONS: Gestational Diabetes
Keywords: Gestational Diabetes; Screening; Cost-effectiveness; obstetrical outcomes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Diabetes in pregnancy or gestational diabetes (GDM) is a condition that, if left untreated, may lead to complications for the mother and her baby. It is still not known which is the best method to diagnosis GDM. The goal of this study is to compare three well-accepted methods for diagnosis of GDM (using either 75 g or 100 g in the glucose tolerance test) and determine which method is the easiest and least expensive to use in relation to the reference method used over the last 20 years. The goal is to see if they can equally predict the healthy outcome of the pregnant mother and her newborn.

DETAILED DESCRIPTION:
Title: What is the optimal method for screening and diagnosis of gestational diabetes? A randomised clinical trial to evaluate incidence of GDM, cost-effectiveness and clinical outcomes using three methods.

Objectives: 1) To evaluate the incidence and cost-effectiveness of screening and diagnosis of GDM by comparing three different methods. 2) To evaluate the following by each method: population characteristics; gestational age at screening, diagnosis and initiation of treatment; and maternal and neonatal outcomes.

Rationale: There is no consensus on the best method to identify cases of GDM, numerous screening and diagnostic procedures are employed worldwide. Recently the Canadian Guidelines recommended a new set of values based on normative data, yet these data have not been validated against a large population and compared with diagnostic rates and outcomes head to head against the long accepted values of O'Sullivan and Mahan. In addition, the question of cost in a Canadian healthcare setting has never been addressed yet it is a significant societal concern. The results of this study would help clarify these issues using evidence-based methodology.

Outline: Pregnant women referred as outpatients for glucose testing for GDM will be given a study information sheet by obstetrics staff. At the time of booking the test they will be reminded of the study and to arrive fasting. On the day of glucose testing, the research assistant will invite patients to participate, obtain consent and perform randomisation into one three groups:

(1) 50g screen ± 100g 3h GTT; (2) 50g screen ± 75g 2h GTT; or (3) 75g 2h GTT. During the glucose test, study participants will also be asked information on health and costs incurred for the process of glucose testing. If the screen or GTT needs to be repeated at some time during the pregnancy, patients will remain in the same study arm as originally assigned. Interpretation of results by patient's caregivers and referral to the diabetes clinic as needed will continue as usual. Data will be analysed using appropriate bivariate and multivariate methods for GDM incidence, direct and indirect costs of glucose testing, and maternal and infant outcomes.

Significance to DM: This study will evaluate the diagnostic efficacy, cost-effectiveness and clinical outcomes of three methods. A one-step procedure may be better tolerated compared to a two-step approach with respect to number of visits, amount of drink and length of testing. Furthermore, diagnosis by a single test may avoid unnecessary delay in initiation of therapy and still identify those patients at risk for type 2 DM.

ELIGIBILITY:
Inclusion Criteria:

* all women presenting for glucose screening in pregnancy between January 2001 and June, 2004 at a tertiary care university hospital setting

Exclusion Criteria:

* insufficient knowledge of French or English; known diabetes; refusal to participate; error in protocol; not fasting when presenting for study test

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5800
Dates: Start 2001-01; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Sara J Meltzer, MD, FRCPC, Principal Investigator — McGill Unversity, Faculty of Medicine, Dept. of Medicine and Obstetrics and Gynecology
Locations (1):
- Royal Victoria Hospital, McGill University Health Centre, Montreal, Quebec, Canada